CLINICAL TRIAL: NCT01307527
Title: Riboflavin Corneal Crosslinking for Brittle Cornea Syndrome and Ehlers-Danlos Syndrome Type VI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Joshua Kruger, Hadassah Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BTL-CXL-HMO-CTIL
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-02

CONDITIONS: Brittle Cornea Syndrome; Ehlers-Danlos Syndrome Type 6
MeSH Terms: conditions — Brittle cornea syndrome 1; Ehlers-Danlos syndrome type 6 | interventions — Riboflavin

INTERVENTIONS:
Drug: Riboflavin — 0.1%, applied every 5 minutes for 60 minutes
Device: Kera-X — 3 mW/cm2, to the central 7.5 mm of the cornea, for 30 minutes

SUMMARY:
Brittle Cornea Syndrome and Ehlers-Danlos Syndrome (EDS) type VI are rare collagen-connective tissue disorders that predispose affected individuals to the development of perforated corneas from the mildest of eye trauma or even spontaneously. Clinical studies evaluating riboflavin-corneal crosslinking have found that it dramatically increases corneal rigidity. Given the success and safety of riboflavin crosslinking, the investigators believe that it can increase the corneal stability in patients affected these disseases, preventing perforation. It is furthermore possible, that riboflavin crosslinking will allow corneal transplants to successfully be performed on blind eyes that have already perforated and opacified. The purpose of the study is to determine whether corneal crosslinking can be safely performed on individuals with Brittle Cornea Syndrome or Ehlers-Danlos Syndrome type VI.

ELIGIBILITY:
Inclusion Criteria:

Adult Patient with:

1. Genetic diagnosis of either Brittle Cornea Syndrome or EDS-VI, and
2. Either:

   * Personal History of either spontaneous corneal perforation or corneal perforation due to minor ocular mechanical trauma or
   * Immediate family member with history of either spontaneous corneal perforation or corneal perforation due to minor ocular mechanical trauma

Exclusion Criteria:

* Any patient that is deemed to be unable to fully cooperate during the crosslinking procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)

PRIMARY OUTCOMES:
Adverse Events from Cornea Riboflavin Crosslinking in Brittle Cornea Syndrome or Ehlers Danlos Type VI | 3 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel